CLINICAL TRIAL: NCT03513172
Title: Hypotensive Efficacy of Topical Prophylaxis for Intraocular Pressure Spikes Following Intravitreal Injections of Anti-vascular Endothelial Growth Factor Agents
Brief Title: Pre-Administration of Brimonidine in Intravitreal Anti-VEGF Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Dr. Efrem Mandelcorn (Unknown)
Responsible Party: Principal Investigator, Tina Felfeli, Medical Student, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 15-9762-B
Record Dates: First submitted 2018-04-17; First posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Post-Injection Intraocular Pressure Spikes
Keywords: Intraocular Pressure; Anti-VEGF Agents; alpha2-agonists
MeSH Terms: interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brimonidine Pre-Administration During First Visit (Active Comparator)
  Interventions: Drug: topical brimonidine tartrate 0.15% (Alphagan® P; Allergan, Inc)
- Brimonidine Pre-Administration During Second Visit (Active Comparator)
  Interventions: Drug: topical brimonidine tartrate 0.15% (Alphagan® P; Allergan, Inc)

INTERVENTIONS:
Drug: topical brimonidine tartrate 0.15% (Alphagan® P; Allergan, Inc) — The rapid hypotensive effects of topical alpha2-agonists such as brimonidine tartrate on decreasing aqueous production and increasing uveoscleral outflow, in addition to their neuroprotective properties, make them an attractive option for prophylactic treatment of post-injection IOP spikes.

SUMMARY:
In this study, investigators will be examining the intraocular pressure lowering effect of brimonidine 0.15% when administered 20min prior to intravitreal anti-VEGF injection.

DETAILED DESCRIPTION:
A total of 55 consecutive patients undergoing anti-VEGF intravitreal injections (received ≥1 treatments) for age-related macular degeneration (AMD), diabetic macular edema (DME) or macula edema secondary to branch retinal vein occlusion (BRVO) will be prospectively recruited between December 2016 and July 2017. Patients will be randomly assigned based on a pre-determined allocation sequence to receive topical brimonidine tartrate 0.15% (Alphagan® P; Allergan, Inc) during either the first or second of two consecutive visits. A standard protocol for sterile preparation with topical 5% povidone-iodine solution will be followed. Pre-injection IOP measurements will be recorded prior to the instillation of dilating agents and brimonidine tartrate. A total of three IOP measurements will be taken by certified ophthalmic technicians at immediately after the injection (T0), 10 minutes after (T10) and 20 minutes after (T20) injection.

ELIGIBILITY:
Inclusion Criteria:

* received ≥1 treatments for age-related macular degeneration (AMD), diabetic macular edema (DME) or macula edema secondary to branch retinal vein occlusion (BRVO)

Exclusion Criteria:

* baseline diagnosis of glaucoma
* baseline IOP during last visit of greater than 21 mmHg
* ongoing use of topical medications (eg. corticosteroids)
* pseudophakic with an anterior chamber intraocular lens
* history of ocular conditions that may impact IOP (eg. pseudoexfoliation)
* previous in-office (eg. laser peripheral iridotomy) and vitreoretinal surgical procedures (eg. pars plana vitrectomy).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Post-Injection Intraocular Pressure Spike | Change from immediately, 10 minutes and 20 minutes after injection
  the intraocular pressure lowering effect of brimonidine 0.15% ophthalmic eye drop when administered 20 minutes prior to intravitreal anti-VEGF injection

CONTACTS AND LOCATIONS:
Overall Officials: Efrem Mandelcorn, MD, FRCSC, Principal Investigator — University Health Network, Toronto

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kampougeris G, Spyropoulos D, Mitropoulou A. Intraocular Pressure rise after Anti-VEGF Treatment: Prevalence, Possible Mechanisms and Correlations. J Curr Glaucoma Pract. 2013 Jan-Apr;7(1):19-24. doi: 10.5005/jp-journals-10008-1132. Epub 2013 Jan 15. PMID 26997776
- [Background] Kim YJ, Sung KR, Lee KS, Joe SG, Lee JY, Kim JG, Yoon YH. Long-term effects of multiple intravitreal antivascular endothelial growth factor injections on intraocular pressure. Am J Ophthalmol. 2014 Jun;157(6):1266-1271.e1. doi: 10.1016/j.ajo.2014.02.035. Epub 2014 Feb 18. PMID 24561173
- [Background] Hoang QV, Mendonca LS, Della Torre KE, Jung JJ, Tsuang AJ, Freund KB. Effect on intraocular pressure in patients receiving unilateral intravitreal anti-vascular endothelial growth factor injections. Ophthalmology. 2012 Feb;119(2):321-6. doi: 10.1016/j.ophtha.2011.08.011. Epub 2011 Nov 4. PMID 22054994
- [Background] Tseng JJ, Vance SK, Della Torre KE, Mendonca LS, Cooney MJ, Klancnik JM, Sorenson JA, Freund KB. Sustained increased intraocular pressure related to intravitreal antivascular endothelial growth factor therapy for neovascular age-related macular degeneration. J Glaucoma. 2012 Apr-May;21(4):241-7. doi: 10.1097/IJG.0b013e31820d7d19. PMID 21423038
- [Background] Aref AA. Management of immediate and sustained intraocular pressure rise associated with intravitreal antivascular endothelial growth factor injection therapy. Curr Opin Ophthalmol. 2012 Mar;23(2):105-10. doi: 10.1097/ICU.0b013e32834ff41d. PMID 22249237
- [Derived] Felfeli T, Hostovsky A, Trussart R, Yan P, Brent MH, Mandelcorn ED. Hypotensive efficacy of topical brimonidine for intraocular pressure spikes following intravitreal injections of antivascular endothelial growth factor agents: a randomised crossover trial. Br J Ophthalmol. 2019 Oct;103(10):1388-1394. doi: 10.1136/bjophthalmol-2018-312603. Epub 2018 Dec 20. PMID 30573499